CLINICAL TRIAL: NCT00529165
Title: The Necessity of an Injection-Meal-Interval in Patients With Type 2 Diabetes Mellitus and Therapy With Human Insulin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jena (Other)
Responsible Party: Prof. Dr. med. Ulrich Alfons Müller, University Hospital Jena
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ISRCTN04277490
Record Dates: First submitted 2007-09-13; First posted 2007-09-14 (Estimated); Last update posted 2009-01-14 (Estimated); Status verified 2009-01

CONDITIONS: Diabetes Mellitus Type 2
Keywords: injection to meal time; human insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): with injection-meal-interval,cross over after 3 month, than without injection-meal-interval for 3 month
  Interventions: Procedure: injection-meal-interval
- B (Experimental): without injection-meal-interval,cross over after 3 month, than with injection-meal-interval for 3 month
  Interventions: Procedure: injection-meal-interval

INTERVENTIONS:
Procedure: injection-meal-interval — The patient injects human insulin (as Actrapid from NovoNordisc) as usual in their insulin routine. The injection is subcutaneous and the dosage is dependent on the blood glucose monitoring. Patients will inject insulin previous every meal, with the following differences:
  1. Group A: with injection-meal-interval: 50 patients educated to inject the insulin with an injection-meal-interval of 15 minutes
  2. Group B: without injection-meal-interval: 50 patients educated to inject the insulin without injection-meal-interval
  Cross-over will occur to the other group after 12 weeks. The follow up is 28 weeks.

SUMMARY:
The purpose of the study is to demonstrate, that there is no difference in metabolic control in patients with type 2 diabetes mellitus and therapy with human insulin with or without injection-meal-interval.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* Aged 40 - 80 years
* Therapy with human insulin

Exclusion Criteria:

* Pregnancy
* Nutrition disorders
* Psychological disease
* Body Mass Index (BMI) less than 25 kg/m^2
* HbA1c greater than 9%

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-07; Primary Completion 2008-07 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
HbA1c | Week 16 and 28

SECONDARY OUTCOMES:
Hypoglycemia | Week 16 and 28
Treatment satisfaction | week 16 and 28
Quality of Life | week 16 and 28

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich A Mueller, Professor, Principal Investigator — University of Jena, department of internal medicine III
Locations (1):
- Friedrich-Schiller-University, department of internal medicine III, Jena, Germany

REFERENCES:
- [Derived] Muller N, Frank T, Kloos C, Lehmann T, Wolf G, Muller UA. Randomized crossover study to examine the necessity of an injection-to-meal interval in patients with type 2 diabetes and human insulin. Diabetes Care. 2013 Jul;36(7):1865-9. doi: 10.2337/dc12-1694. Epub 2013 Jan 22. PMID 23340895
- [Derived] Muller N, Kloos C, Frank T, Ristow M, Wolf G, Muller UA. Prevalence of injection-meal interval usage and its association with variables of metabolic control in patients with Type 1 and Type 2 diabetes. Diabet Med. 2011 Feb;28(2):223-6. doi: 10.1111/j.1464-5491.2010.03172.x. PMID 21219434